CLINICAL TRIAL: NCT06691542
Title: Efficacy and Safety of Platelet-rich Plasma, Metformin and Cryotherapy in Treatment of Non-genital Warts
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Gamal Abd El-Wahab Mahmoud, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP, Metformin in warts
Record Dates: First submitted 2024-02-09; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Non-Genital Warts
MeSH Terms: interventions — Metformin; Cryotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intralesional injection of Metformin (Experimental): Group 1: will include 36 patients with multiple common, plantar and/or plane warts. They will be treated by intralesional injection of metformin using insulin syringe every 2-weeks until complete clearance or for a maximum of 6 sessions.
  Interventions: Drug: Metformin
- Intralesional injection of platelet- rich plasma (Experimental): Group 2: will include 36 patients with multiple common, plantar and/or plane warts. They will be treated by intralesional injection of platelet- rich plasma into the warts by an insulin syringe every 2 weeks until complete clearance or for a maximum of 6 sessions
  Interventions: Drug: platelet-rich plasma
- Cryotherapy (Experimental): Group 3: will include 36 patients with multiple common, plantar and/or plane warts. They will receive cryotherapy sessions every two weeks until complete clearance or for a maximum of 6 sessions.
  Interventions: Other: cryotherapy

INTERVENTIONS:
Drug: platelet-rich plasma — platelet-rich plasma, metformin and cryotherapy in treatment of non-genital warts
  Arms: Intralesional injection of platelet- rich plasma
Drug: Metformin — platelet-rich plasma, metformin and cryotherapy in treatment of non-genital warts
  Arms: Intralesional injection of Metformin
Other: cryotherapy — platelet-rich plasma, metformin and cryotherapy in treatment of non-genital warts
  Arms: Cryotherapy

SUMMARY:
1. Evaluation of the efficacy and safety of intralesional injection of autologous platelet-rich plasma in treatment of various types of cutaneous non genital warts
2. Evaluation of the efficacy and safety of intralesional injection of metformin in treatment of various types of cutaneous non genital warts
3. Comparing the efficacy and safety of intralesional injection of autologous platelet-rich plasma and intralesional injection of metformin with that of cryocautery in treatment of various types of cutaneous non genital warts.

DETAILED DESCRIPTION:
Cutaneous warts caused by human papillomavirus (HPV) are benign proliferative lesions that occur at any age in human life.

More than 100 different types of HPVs have been fully characterized . Warts may exist in different forms according to the epithelial surface affected and HPV type responsible for the infection. Common warts (Verruca vulgaris), plantar warts (Verruca plantaris), flat or plane warts (Verruca plana) and genital warts (Condyloma acuminata) are some of the clinical manifestations of HPV infection .

Although lesions can resolve spontaneously within 2 years without treatment, treatment is sought by many who are unwilling to wait for spontaneous clearance, by those who do not experience such resolution and for reasons of preventing infections of other individuals and reducing the risk of malignancy . Additionally, pain, discomfort, recurrent bleeding, functional limitation, and esthetic disfigurements due to cutaneous warts are common indications for seeking treatment.

Several therapeutic modalities have been used to treat HPV infections. The choice of treatment should take into account factors such as age, location, number and size of the lesions, clinical subtype and the patient's immunological status.

Available treatments are aimed at either breakdown or removal of visible warts or induction of cytotoxicity against infected cells .

They include destructive agents (keratolytic, cryotherapy, curettage and cautery, laser, photodynamic therapy), antimitotic agents (podophyllin, bleomycin, retinoids), immune stimulants (topical sensitizers, cimetidine), and topical virucidal agents [formaldehyde (formalin), glutaraldehyde (Glutaral) .

Unfortunately, no single treatment is satisfactory for all patients. Many treatments are time consuming, painful and can leave scars or hypopigmentation; moreover, recurrence rates after any treatment range from 6% to 100% . So, the development of new effective and safe treatments seems to be an urgent need.

Cryocautery represents a first line of therapy for cutaneous warts. It uses liquid nitrogen to freeze tissues and destroy warts.

Liquid nitrogen cryotherapy involves freezing a wart with liquid nitrogen for 10 to 20 seconds every two to three weeks. Precisely how cryotherapy destroys warts is not well understood, but the prevailing theory is that freezing causes local irritation, leading the host to mount an immune reaction against the virus.

However, side effects for cryocautery are common, they include pain, depigmentation, delayed healing, ulceration, scar formation and recurrence

Platelet- rich plasma (PRP) is a small volume of plasma rich in platelets. It has become a hopeful therapy in the last decade to treat several cutaneous diseases due to its increased concentrations of growth factors. As it is of autologous origin, it reduces the possibility of adverse effects and transfusion transmitted infections.

PRP has been utilized in the treatment of numerous cutaneous diseases such as alopecia, skin ulcers, and acne vulgaris. Its utility has been extended to other cutaneous diseases as melasma, hyperpigmentation, and burns, in addition to its usefulness in tissue repair and regeneration.

To the best of our knowledge the efficacy of PRP in the treatment of plane warts was assessed in a single uncontrolled clinical trial which revealed that intralesional injection of PRP was effective and well-tolerated immunotherapy for treating of multiple recalcitrant plane warts.

Moreover, complete remission of multiple resistant plantar warts after treatment by combined intralesional autologous PRP injections and local application of salicylic acid 30% was observed in only one case report.

Mechanisms suggested for such promising response of warts to intralesional injection of PRP included induction of expression of numerous pro-inflammatory cytokines as interleukin-6, interleukin-8, tumor necrosis factor-alpha, and C-C motif chemokine ligand 5 which then activate several immune cells leading to increased inflammation.

Also, platelets expressed CD40L, on its activation; it modulates its interaction with CD40 presenting on macrophages, B-cells, monocytes, endothelial cells, dendritic cells, and mediates their activities.

Platelets may modulate the innate immunity and provide antimicrobial activities either by synthesis of antimicrobial peptides or by modulating the immune activities of other immune cells as neutrophils and monocytes.

These interesting findings open the way for future studies to evaluate the usefulness of PRP in treating different clinical types of warts.

Metformin, a widely used drug to treat type 2 diabetes mellitus and metabolic syndrome, has been used systemically in different dermatological diseases such as hormonal acne, hidradenitis suppurativa (HS) and acanthosis nigricans in which it may act through improving hyperinsulinemia . Additionally, it was found effective when used topically in treatment of melasma with an equivalent effect to triple combination cream , and acne vulgaris .

Metformin has immunomodulatory activity that reduces the production of proinflammatory cytokines, it also inhibits the cytokine production of pathogenic Th1 and Th17 cells .

Furthermore, many studies, both in vitro and in vivo with small animal models, have highlighted the antiviral properties of metformin.

Additionally, Metformin has shown antitumorigenic potential in HPV-positive cancer cells. Such properties suggests that metformin might be effective therapeutic option for viral warts. However, to the best of our knowledge, no studies have been conducted to explore that hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cutaneous (extragenital) viral warts (single , new or recurrent, common, plane and/or planter warts.
* Age ranged from 8 to 60 years old.
* No concurrent systemic or topical treatment of warts.

Exclusion Criteria:

* Patients with fever or signs of any inflammation or infection
* Pregnancy and lactation.
* Immunosuppression or being under any kind of treatment causing absolute or relative immunosuppression.
* History of any bleeding, clotting disorder or using anticoagulants
* Chronic systemic diseases such as diabetes, chronic renal failure, hepatic insufficiency, and cardiovascular disorders.
* atients using concurrent treatments for warts or one month before .
* Any generalized dermatitis, allergic skin disorders

Ages: 8 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-11-14 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Complete resolution of the wart(s) by disappearance of the wart and return of the normal skin markings | 3 months
  Complete resolution of the wart(s) by disappearance of the wart and return of the normal skin markings

SECONDARY OUTCOMES:
•Change in size in millemeter | 3 months
  Change in size in millemeter
•Decrease in numbers of the warts | 3 months
  Decrease in numbers of the warts
•Recurrence rates at 3 months for wart(s) with complete resolution. | 3 months
  Recurrence rates at 3 months for wart(s) with complete resolution.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Mohamed Kamal Elsayed Youssef, prof, Principal Investigator — Professor of Dermatology and Venereology Faculty of Medicine, Assiut University; Alaa Mohamed Mahmoud Hamdy Ghazally, Lecturer, Principal Investigator — Lecturer of Dermatology and Venereology Faculty of Medicine, Assiut University

REFERENCES:
- [Background] Zhu P, Qi RQ, Yang Y, Huo W, Zhang Y, He L, Wang G, Xu J, Zhang F, Yang R, Tu P, Ma L, Liu Q, Li Y, Gu H, Cheng B, Chen X, Chen A, Xiao S, Jin H, Zhang J, Li S, Yao Z, Pan W, Yang H, Shen Z, Cheng H, Song P, Fu L, Chen H, Geng S, Zeng K, Wang J, Tao J, Chen Y, Wang X, Gao XH. Clinical guideline for the diagnosis and treatment of cutaneous warts (2022). J Evid Based Med. 2022 Sep;15(3):284-301. doi: 10.1111/jebm.12494. Epub 2022 Sep 18. PMID 36117295
- [Background] Araujo MG, Magalhaes GM, Garcia LC, Vieira EC, Carvalho-Leite MLR, Guedes ACM. Update on human papillomavirus - Part II: complementary diagnosis, treatment and prophylaxis. An Bras Dermatol. 2021 Mar-Apr;96(2):125-138. doi: 10.1016/j.abd.2020.11.005. Epub 2021 Feb 16. PMID 33637397
- [Background] Sterling JC, Gibbs S, Haque Hussain SS, Mohd Mustapa MF, Handfield-Jones SE. British Association of Dermatologists' guidelines for the management of cutaneous warts 2014. Br J Dermatol. 2014 Oct;171(4):696-712. doi: 10.1111/bjd.13310. Epub 2014 Oct 1. No abstract available. PMID 25273231
- [Background] Bacelieri R, Johnson SM. Cutaneous warts: an evidence-based approach to therapy. Am Fam Physician. 2005 Aug 15;72(4):647-52. PMID 16127954
- [Background] Focht DR 3rd, Spicer C, Fairchok MP. The efficacy of duct tape vs cryotherapy in the treatment of verruca vulgaris (the common wart). Arch Pediatr Adolesc Med. 2002 Oct;156(10):971-4. doi: 10.1001/archpedi.156.10.971. PMID 12361440
- [Background] Abu El-Hamd M, Aboeldahab S. Possible clinical efficacy and tolerability of platelet-rich plasma in the treatment of patients with recalcitrant plane warts: The first clinical study. J Cosmet Dermatol. 2021 Nov;20(11):3623-3629. doi: 10.1111/jocd.14008. Epub 2021 Mar 1. PMID 33599062
- [Background] Abu El-Hamd M, Aboeldahab S. A case of resistant multiple plantar warts cured with combined autologous platelet-rich plasma injection and topical salicylic acid 30. J Cosmet Dermatol. 2022 Jun;21(6):2417-2419. doi: 10.1111/jocd.14468. Epub 2021 Sep 24. PMID 34559938
- [Background] McDonald B, Dunbar M. Platelets and Intravascular Immunity: Guardians of the Vascular Space During Bloodstream Infections and Sepsis. Front Immunol. 2019 Oct 11;10:2400. doi: 10.3389/fimmu.2019.02400. eCollection 2019. PMID 31681291
- [Background] Henn V, Slupsky JR, Grafe M, Anagnostopoulos I, Forster R, Muller-Berghaus G, Kroczek RA. CD40 ligand on activated platelets triggers an inflammatory reaction of endothelial cells. Nature. 1998 Feb 5;391(6667):591-4. doi: 10.1038/35393. PMID 9468137
- [Background] Flad HD, Brandt E. Platelet-derived chemokines: pathophysiology and therapeutic aspects. Cell Mol Life Sci. 2010 Jul;67(14):2363-86. doi: 10.1007/s00018-010-0306-x. Epub 2010 Mar 7. PMID 20213276
- [Background] Chen X, Guo H, Qiu L, Zhang C, Deng Q, Leng Q. Immunomodulatory and Antiviral Activity of Metformin and Its Potential Implications in Treating Coronavirus Disease 2019 and Lung Injury. Front Immunol. 2020 Aug 18;11:2056. doi: 10.3389/fimmu.2020.02056. eCollection 2020. PMID 32973814
- [Background] Benedetti F, Sorrenti V, Buriani A, Fortinguerra S, Scapagnini G, Zella D. Resveratrol, Rapamycin and Metformin as Modulators of Antiviral Pathways. Viruses. 2020 Dec 17;12(12):1458. doi: 10.3390/v12121458. PMID 33348714
- [Background] Hoppe-Seyler K, Herrmann AL, Daschle A, Kuhn BJ, Strobel TD, Lohrey C, Bulkescher J, Krijgsveld J, Hoppe-Seyler F. Effects of Metformin on the virus/host cell crosstalk in human papillomavirus-positive cancer cells. Int J Cancer. 2021 Sep 1;149(5):1137-1149. doi: 10.1002/ijc.33594. Epub 2021 May 6. PMID 33844847
- [Background] Abou-Taleb DAE, Abou-Taleb HA, El-Badawy O, Ahmed AO, Thabiet Hassan AE, Awad SM. Intralesional vitamin D3 versus intralesional purified protein derivative in treatment of multiple warts: A comparative clinical and immunological study. Dermatol Ther. 2019 Sep;32(5):e13034. doi: 10.1111/dth.13034. Epub 2019 Aug 7. PMID 31355514
- [Background] Abd El-Magiud EM, Abd El-Samea GM, Gaber HD. Intralesional injection of measles, mumps, and rubella vaccine versus cryotherapy in treatment of warts: A randomized controlled trial. Dermatol Ther. 2020 Mar;33(2):e13257. doi: 10.1111/dth.13257. Epub 2020 Feb 16. PMID 32031726